CLINICAL TRIAL: NCT01224847
Title: Intravitreal Injection Anesthesia - Comparison of Different Topical Agents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Thomas G. Sheidow, MD, FRCSC, Ophthalmologist, Vitreoretinal Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R-09-415; 16454 (Other: REB)
Record Dates: First submitted 2010-10-06; First posted 2010-10-20 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Age-Related Macular Degeneration (AMD)
Keywords: AMD; Intravitreal Injection; Anesthesia
MeSH Terms: conditions — Macular Degeneration | interventions — Tetracaine; Cocaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tetracaine gtt (Active Comparator): Pre-Intravitreal injection - 1 gtt Tetracaine topically
  Interventions: Drug: Tetracaine
- Tetraciane gtt + Lidocaine pledget (Active Comparator): 1 gtt Tetracaine pre-IVT injection + application Lidocaine pledget to injection site
  Interventions: Drug: Lidocaine
- Cocaine gtt alone (Active Comparator): 1 gtt pre-IVT injection
  Interventions: Drug: Cocaine

INTERVENTIONS:
Drug: Tetracaine — 1 gtt
  Arms: Tetracaine gtt
Drug: Cocaine — 1 gtt
  Arms: Cocaine gtt alone
Drug: Lidocaine — Lidocaine soaked pledget
  Arms: Tetraciane gtt + Lidocaine pledget

SUMMARY:
Patients with neovascular age-related macular degeneration (AMD) scheduled to receive intravitreal (IVT) Ranibizumab injection will be randomized to receive one of three topical anesthetics: (1) tetracaine drop (gtt) + lidocaine pledget to the injection site for 10 seconds (2) tetracaine gtt alone and (3) cocaine gtt alone. A questionnaire will be conducted immediately after and 15 minutes after the injection, to assess for pain.

DETAILED DESCRIPTION:
All patients scheduled to receive intravitreal Ranibizumab for the treatment of neovascular AMD will be evaluated for inclusion into the study. After a positive evaluation, the study will be explained to the patient, the Letter of Explanation reviewed with the patient and informed consent approved if patient agrees to participate. Demographic data of sex and age will be recorded. As well the number of previous intravitreal injections will be recorded ( none, 2 - 5 and > 5 ). A nurse will then proceed to select an opaque envelope from a box of identical envelopes. The envelope will contain the topical anesthetic agent to be used. The randomization code linking each patient to their anesthetic will be stored in a secure location, and only accessed at the completion of the trial. The anesthetic procedure will be performed by someone other than the surgeon who will perform the IVT injection. After a minute of the anesthetic application, the surgeon, blinded to the anesthetic intervention, will perform the IVT injection of Ranibizumab. Immediately following the injection, a blinded observer will first explain the Pain Questionnaire, and then conduct it. Also at this time, the physician who performed the injection will complete the Wong-Baker Pain Questionnaire. The patient will then be asked to wait in a room for an additional 15 minutes, where the same observer will return and the Pain Questionnaire will be conducted a second time.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 50
2. Scheduled to receive Ranibizumab for neovascular AMD

Exclusion Criteria:

1. History of pars plana vitrectomy
2. Any major surgery within the prior 28 days, or one planned within next 6 months
3. History of thromboembolic event
4. Previous known allergic response to topical anesthetic(s) (lidocaine, tetracaine, cocaine)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To elucidate the most effective topical agent for intravitreal injections. | Pain scores reported immediately after intravitreal injection.
  Patients will measure pain by the use of a Visual Analog Scale.

SECONDARY OUTCOMES:
To elucidate the most effective topical agent for intravitreal injections. | Pain scores reported 15 minutes after intravitreal injection.
  Patients will measure pain by the use of a Visual Analog Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Sheidow, MD, FRCSC, Principal Investigator — Ivey Eye Institute, St. Joseph's Health Care
Locations (1):
- Ivey Eye Institute, London, Ontario, Canada